CLINICAL TRIAL: NCT05313412
Title: Clinical Evaluation of Two Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C21-706 (EX-MKTG-127)
Record Dates: First submitted 2022-03-24; First posted 2022-04-06 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, Then Lens B (Experimental): Participants will wear Lens A for six hours and then cross over to wear Lens B for six hours.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)
- Lens B, Then Lens A (Experimental): Participants will wear Lens B for six hours and then cross over to wear Lens A for six hours.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)

INTERVENTIONS:
Device: Lens A (comfilcon A lens) — 6 hours
Device: Lens B (lehfilcon A lens) — 6 hours

SUMMARY:
This study is to compare the short-term clinical performance and subjective acceptance of two silicone hydrogel soft contact lenses.

DETAILED DESCRIPTION:
This is a double-masked, randomized, bilateral crossover study to compare the short-term clinical performance of two silicone hydrogel soft contact lenses. Each lens type is worn for approximately six hours on separate study days, in random sequence.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged between 18 and 40 years.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They have successfully worn contact lenses within six months of starting the study.
5. They can be satisfactorily fitted with the study contact lenses.
6. They have a contact lens spherical prescription between -0.25 to - 6.00D (inclusive) based on the ocular refraction.
7. They have a spectacle cylindrical correction of -0.75D or less in each eye based on the ocular refraction.
8. They own and habitually wear single vision spectacles.
9. They can attain at least 0.20 logMAR distance high contrast visual acuity in each eye, with the study lenses.
10. They agree not to participate in other clinical research while enrolled on this study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contraindicate contact lens wear.
2. They have a systemic disorder which would normally contraindicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (eg HIV) or a history of anaphylaxis or severe allergic reaction.
9. They have grade 3 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality, which would normally contraindicate contact lens wear.
10. They have taken part in any other clinical trial or research, within two weeks prior to starting this study, which may impact on this particular work.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD,MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-eight participants attended the initial visit with all participants completing the study.
Groups:
- Lens A, Then Lens B: Participants wore Lens A for 6 hours and then wore Lens B for 6 hours on two separate study days.
- Lens B, Then Lens A: Participants wore Lens B for 6 hours and then wore Lens A for 6 hours on two separate study days.
Period: Overall Study
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total study population
Arm/Group | Overall Study
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ease of Lens Insertion
Description: Ease of Lens Insertion is measured on a scale of 0-100 (0-Unmanageable, Lenses impossible to insert; 100-Excellent. No problems with lens insertion)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants wore Lens A for six hours.
- Lens B: Participants wore Lens B for six hours.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 38 | 38
units on a scale | 92.1 (10.3) | 90.9 (17.4)

ADVERSE EVENTS:
Time Frame: From dispense up to six hours on each lens type, for a total of 12 hours
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT05313412/Prot_SAP_000.pdf